CLINICAL TRIAL: NCT02187172
Title: A PHASE IV, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY OF THE EFFECTS OF USTEKINUMAB ON VASCULAR INFLAMMATION IN PSORIASIS
Brief Title: Vascular Inflammation in Psoriasis-Ustekinumab (VIP-U)
Acronym: VIP-U
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 820124
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Psoriasis; Cardiovascular Disease
Keywords: Psoriasis; Cardiovascular Disease; Vascular Inflammation; Lipid Biomarkers; FDG-PET/CT
MeSH Terms: conditions — Psoriasis; Cardiovascular Diseases | interventions — Ustekinumab

STUDY DESIGN:
Intervention Model Description: A hybrid RCT (randomized controlled trial) crossover trial where all patients receive total of 52 weeks of active treatment following an RCT phase of 12 weeks (active treatment or placebo). Patients randomized to active treatment will receive additional 40 weeks of active treatment at end of RCT phase; patients randomized to placebo will receive 52 weeks of active treatment at end of RCT phase. Primary outcomes are assessed at end of the RCT phase (comparison of interventions in change from start of treatment) and at end of 52 weeks of active treatment (change from start of treatment).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ustekinumab (Stelara) (Active Comparator): Ustekinumab (Stelara) subcutaneous injection 45mg (if person's weight is 100kg or less) or 90mg (if person's weight is greater than 100kg) at day 0 and week 4 followed by every 12-week dosing thereafter. Patient will receive total of 52 weeks of ustekinumab (12 weeks during RCT phase, 40 weeks post RCT phase). The end of study is at Week 52 for this arm.
  Interventions: Drug: Ustekinumab
- Placebo (Placebo Comparator): Placebo subcutaneous injection will be given according to the same dose and schedule as the active comparator until week 12 (end of RCT phase). At week 12, ustekinumab will be administered according according to the same injection schedule as the active comparator arm for 52 weeks. Patient will receive total of 52 weeks of ustekinumab (0 weeks during RCT phase, 52 weeks post RCT phase). The end of study is at Week 64 for this arm.
  Interventions: Drug: Ustekinumab; Drug: Placebo

INTERVENTIONS:
Drug: Ustekinumab
Drug: Placebo
  Arms: Placebo

SUMMARY:
The VIP-U Study is a clinical trial designed to investigate the effect of ustekinumab (Stelara) and placebo on reducing vascular inflammation and cardiometabolic risk biomarkers in patients with moderate to severe psoriasis.

This study will look for systemic vascular inflammation in study participants with a test called FDG PET/CT (fluorodeoxyglucose-positron emission tomography/computed tomography). The study will also look for cardiometabolic identifiers (heart disease and metabolic factors) in blood samples, including markers of high cholesterol, cholesterol efflux function (the ability of cholesterol to move in the body), metabolic factors, and inflammation.

The study will also examine the effects of ustekinumab compared to placebo on psoriasis activity, severity and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age and older.
2. Clinical diagnosis of psoriasis for at least 6 months as determined by subject interview of his/her medical history and confirmation of diagnosis through physical examination by Investigator.
3. Stable plaque psoriasis for at least 2 months before Screening and at Baseline (Week 0) as determined by subject interview of his/her medical history.
4. Moderate to severe psoriasis defined by ≥ 10 percent Body Surface Area (BSA) involvement at the Baseline (Week 0) visit.
5. PASI score of ≥ 12 at the Baseline (Week 0) visit.
6. Subject is a candidate for systemic therapy and has active psoriasis despite prior treatment with topical agents.
7. Women are eligible to participate in the study if they meet one of the following criteria:

   1. Women of childbearing potential who are willing to undergo periodic pregnancy testing during the study and agree to use at least one method of contraception throughout the study duration and for at least 15 weeks after the last dose of the study drug are eligible to participate.
   2. Women who are postmenopausal (for at least one year), sterile, or hysterectomized are eligible to participate.
   3. Women who have undergone tubal ligation are eligible to participate.
   4. Women who agree to be sexually abstinent, defined as total abstinence from sexual intercourse, as a form of contraception, are eligible to participate.
8. Men are eligible to participate in the study if they meet one of the following criteria:

   1. Agree to use a proven birth control method during the study and for at least 15 weeks after the last dose of the study drug.
   2. Have a female partner who agrees to use at least one method of contraception throughout the study duration and for at least 15 weeks after the last dose of the study drug.
   3. Have a female partner who is postmenopausal (for at least one year), sterile, or hysterectomized;
   4. Have a female partner who has undergone tubal ligation,
   5. Agree to be sexually abstinent, defined as total abstinence from sexual intercourse, as a form of contraception.
9. Subject is judged to be in good general health as determined by the Principal Investigator based upon the results of medical history, laboratory profile, physical examination, and 12-lead electrocardiogram (ECG) performed at screening.
10. Able and willing to give written informed consent and to comply with requirements of this study protocol.

Exclusion Criteria:

1. Previous adverse event following exposure to an IL-12/IL-23 antagonist that led to discontinuation of therapy and contraindicates future treatment.
2. Previous lack of response to an IL-12/IL-23 antagonist that led to discontinuation of therapy.
3. Diagnosis of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis.
4. Diagnosis of other active skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with evaluation of psoriasis.
5. Cannot avoid UVB phototherapy or Excimer laser for at least 14 days prior to the Baseline (Week 0) visit and during the study.
6. Cannot avoid psoralen-UVA phototherapy for at least 30 days prior to the Baseline (Week 0) visit and during the study.
7. Cannot discontinue systemic therapies for the treatment of psoriasis, or systemic therapies known to improve psoriasis, during the study:

   * Systemic therapies must be discontinued at least 30 days prior to the Baseline (Week 0) visit except for biologics.

     * All biologics, except ustekinumab, must be discontinued for at least 90 days prior to Baseline (Week 0).
     * Any IL-12/IL-23 antagonist (e.g., ustekinumab, briakinumab) must be discontinued for at least 180 days prior to Baseline (Week 0).
   * Investigational agents must be discontinued at least 30 days or 5 half-lives (whichever is longer) prior to the Baseline (Week 0) visit.
8. Subject is taking or requires oral or injectable corticosteroids during the study. Inhaled corticosteroids for stable medical conditions are allowed.
9. Poorly controlled medical condition, such as unstable ischemic heart disease, cerebrovascular accident or myocardial infarction within the prior 6 months, psychiatric disease requiring frequent hospitalization, and any other condition, which, in the opinion of the Investigator, would put the subject at risk by participation in the study.
10. History of diabetes mellitus, type 1 or type 2 with the exception that patients with type 2 diabetes may be enrolled if the duration of diabetes is <10 years and HbA1c is <7.0%.
11. Uncontrolled hypertension, with measured systolic blood pressure >180 mmHg or diastolic blood pressure >90 mmHg
12. Subject has infection or risk factors for severe infections, for example:

    * Positive serology or known history of HIV, hepatitis B or C, or other severe, recurrent, or persistent infections;
    * Excessive immunosuppression or other factors associated with it, including human immunodeficiency virus infection;
    * Active tuberculosis (TB) disease;
    * Evidence of latent TB infection demonstrated by positive Quantiferon-GOLD result; except if prophylactic treatment for TB, as recommended by local guidelines, is initiated prior to administration of study drug or if there is documentation that the subject has received prophylactic treatment for TB within 3 years prior to the first administration of study agent.
    * Any other significant infection requiring hospitalization or intravenous (IV) antibiotics in the month prior to Baseline;
    * Infection requiring treatment with oral or parenteral (other than IV) antibiotics within 14 days prior to Baseline;
    * Subject has received vaccination with Bacille Calmette-Guerin (BCG) within 365 days prior to Screening or will receive BCG vaccination during study participation including up to 12 months after the last dose of the study drug;
    * Subject has received vaccination with a live viral agent 30 days prior to Screening or will require a live vaccination during study participation including up to 3 months after the last dose of study drug.
13. Subject has history of hematological or solid malignancy within the past five years other than successfully treated basal cell carcinoma, non-metastatic cutaneous squamous cell carcinoma or cervical carcinoma in situ.
14. Female subject who is pregnant or breast-feeding or considering becoming pregnant during the study.
15. Male subject who is considering fathering a child during the study.
16. Screening clinical laboratory analyses showing any of the following abnormal results:

    * Hemoglobin (Hgb) < 10 g/dL in females or <12 g/dL in males;
    * White blood cell (WBC) count <2.5 x 109/L

      o Subject can be included if WBC count is <2.5 x 109/L and absolute neutrophil count (ANC) is >1000 cells / mm3.
    * WBC count > 15 x 109/L;
    * Platelet count < 100 x 109/L;
    * Serum creatinine >1.6 mg/dL (>141 µmol/L);
    * Serum aspartate transaminase (AST) or alanine transaminase (ALT) >2.5 upper limits of normal (ULN);
    * Serum total bilirubin ≥2 mg/dL (≥26 µmol/L)
17. Recent history of substance abuse or psychiatric illness that could preclude compliance with the protocol.
18. History of any substance abuse within 365 days of screening visit
19. Alcohol use >14 drinks per week at the screening visit or within 30 days of the screening period
20. If subject is on cholesterol-lowering medication (e.g. statin), dose and form of medication must be stable for 90 days prior to week 0 and remain stable throughout the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-07; Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Gelfand, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ustekinumab: Randomized to receive Ustekinumab (Stelara) from day 0 until week 12 (randomized controlled trial (RCT) phase). Continue to receive ustekinumab for additional 40 weeks for a total of 52 weeks of ustekinumab. The end of study is at Week 52 for this arm.
- Placebo: Randomized to receive Placebo from day 0 until week 12 (RCT phase). Receive ustekinumab from week 12 until week 64 for a total of 52 weeks of ustekinumab. The end of study is at Week 64 for this arm.
Period: Overall Study
Arm/Group | Ustekinumab | Placebo
Started | 22 | 21
RCT Phase Completed (Week 12 for both arms) | 22 | 19
Completed (Received total of 52 weeks of ustekinumab. Week 52 for Ustekinumab arm, Week 64 for Placebo arm.) | 19 | 15
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — Lack of Efficacy | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ustekinumab (Stelara): Ustekinumab (Stelara) subcutaneous injection 45mg (if person's weight is 100kg or less) or 90mg (if person's weight is greater than 100kg) at day 0 and week 4 followed by every 12-week dosing thereafter.
  Ustekinumab
- Placebo: Placebo subcutaneous injection will be given according to the same dose and schedule as the active comparator.
  Ustekinumab
  Placebo
- Total: Total of all reporting groups
Arm/Group | Ustekinumab (Stelara) | Placebo | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.45 (13.6) | 45.33 (12.76) | 42.33 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 19 | 12 | 31
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.24 (7.95) | 33.32 (6.29) | 33.28 (7.1)
Medical History [Number; unit: participants]
  Arthritis | 0 | 1 | 1
  Coronary Artery Disease | 1 | 1 | 2
  Depression | 2 | 2 | 4
  Diabetes | 0 | 1 | 1
  Hyperlipidemia | 5 | 2 | 7
  Stroke | 1 | 0 | 1
  Statin Use | 3 | 3 | 6
Body Surface Area (BSA) [Mean (Standard Deviation); unit: percentage of total body surface area] | 26.18 (17.51) | 23.71 (15.58) | 24.98 (16.45)
Psoriasis Area Severity Index (PASI) score [Mean (Standard Deviation); unit: composite score] — Psoriasis Area and Severity Index (PASI) combines the assessment of the severity of lesions and the area affected into a single score with range 0 (no disease) to 72 maximal disease.
  composite score | 20.03 (7.47) | 19.82 (7.64) | 19.93 (7.46)
Physician Global Assessment (PGA) [Mean (Standard Deviation); unit: calculated score] — The Physician Global Assessment (PGA) is an average assessment of all psoriatic lesions based on erythema, scale, and induration with score range 0 (no disease/clear) to 5 (maximal disease).
  calculated score | 3.5 (0.57) | 3.38 (0.8) | 3.44 (0.69)
Psoriasis duration [Mean (Standard Deviation); unit: years] | 16.45 (11.02) | 20.29 (14.41) | 18.13 (12.58)
Psoriasis treatment history [Number; unit: participants]
  Biologics | 10 | 9 | 19
  Systemics | 6 | 2 | 8
  Phototherapy | 10 | 9 | 19
Psoriatic Arthritis (PsA) present [Count of Participants; unit: Participants] | 1 | 6 | 7
Age at PsA diagnosis [Mean (Standard Deviation); unit: years] — Population: Only applicable in patients with psoriatic arthritis
  years
    number analyzed (Participants) | 1 | 5 | 6
    (all) | 22 (0) | 43.6 (14.33) | 40 (15.56)

OUTCOME MEASURES:

1. Primary Outcome: Change in Vascular Inflammation
Description: Change in total vascular inflammation of five aortic segments as assessed on FDG-PET/CT between baseline and week 12 (RCT period) or end of study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period). The arterial uptake of FDG is measured by the standardized uptake value (SUV) max divided by the venous SUV mean yielding a target to background ratio (TBR).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: The number of subjects analyzed reflect patient dropouts and availability of analyzable samples. The two arms in the RCT period are compared in Statistical Analysis 1. The composite "Total" group is used to assess 52 weeks of active treatment at end of study compared to baseline and is analyzed separately in Statistical Analysis 2.
Measure: Mean (Standard Error); unit: TBR max
Groups:
- Ustekinumab (RCT Period): Randomized to receive Ustekinumab (Stelara) from day 0 until week 12. Outcome measures reflect changes at week 12 compared to baseline.
- Placebo (RCT Period): Randomized to receive Placebo from day 0 until week 12. Outcome measures reflect changes at week 12 compared to baseline.
- Total (Active Treatment Period): Combined ustekinumab and placebo groups for active treatment period analysis. Outcome measures reflect changes at end of study (week 52 for group randomized to Ustekinumab, week 64 for group randomized to Placebo) compared to baseline.
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 22 | 19 | 38
TBR max | -0.1015 (0.0465) | 0.1442 (0.0137) | -0.0151 (0.0353)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0012, Regression, Linear; Mean Difference (Final Values) = -0.2456, 95% CI 2-sided [-0.3873 to -0.1040], Standard Error of Mean 0.0700
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.6718, Regression, Linear; Mean Difference (Final Values) = -0.0151, 95% CI 2-sided [-0.0867 to 0.0565], Standard Error of Mean 0.0353

2. Primary Outcome: Change in Inflammatory Biomarker Levels: Intercellular Adhesion Molecule-1 (ICAM-1)
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on ICAM-1, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
ng/mL | 10.83 (26.30) | 75.80 (37.19) | 6.65 (22.24)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.1159, Regression, Linear; Mean Difference (Final Values) = -64.97, 95% CI 2-sided [-115.83 to 25.89], Standard Error of Mean 44.88
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.7666, Regression, Linear; Mean Difference (Final Values) = 6.65, 95% CI 2-sided [-38.41 to 51.72], Standard Error of Mean 22.24

3. Primary Outcome: Change in Inflammatory Biomarker Levels: Vascular Cell Adhesion Molecule-1 (VCAM-1)
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on VCAM-1, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
ng/mL | -20.36 (18.39) | 60.53 (24.76) | -1.99 (14.11)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0115, Regression, Linear; Mean Difference (Final Values) = -80.89, 95% CI 2-sided [-142.55 to -19.23], Standard Error of Mean 30.46
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.8883, Regression, Linear; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-30.58 to 26.59], Standard Error of Mean 14.11

4. Primary Outcome: Change in Inflammatory Biomarker Levels: C-reactive Protein (CRP)
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on CRP, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
ng/mL | -2886.57 (2851.16) | 140.64 (1108.54) | -1974.63 (1659.11)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.3472, Regression, Linear; Mean Difference (Final Values) = -3027.21, 95% CI 2-sided [-9465.95 to 3411.54], Standard Error of Mean 3180.58
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Combined ustekinumab and placebo groups for active treatment period analysis; Test type: Superiority; p = 0.2416, Regression, Linear; Mean Difference (Final Values) = -1974.63, 95% CI 2-sided [-5336.30 to 1387.04], Standard Error of Mean 1659.11

5. Primary Outcome: Change in Inflammatory Biomarker Levels: Ferritin
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Ferritin, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
ng/mL | -12.32 (39.16) | -32.97 (27.40) | 47.00 (35.84)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.6742, Regression, Linear; Mean Difference (Final Values) = 20.66, 95% CI 2-sided [-78.03 to 119.34], Standard Error of Mean 24.75
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.1979, Regression, Linear; Mean Difference (Final Values) = 47.00, 95% CI 2-sided [-25.63 to 11963], Standard Error of Mean 35.84

6. Primary Outcome: Change in Inflammatory Biomarker Levels: Serum Amyloid A (SAA)
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on SAA, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
ng/mL | -7687.80 (7389.00) | 196.49 (203.34) | -3782.54 (4073.25)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.3173, Regression, Linear; Mean Difference (Final Values) = -7884.29, 95% CI 2-sided [-23634.67 to 7566.10], Standard Error of Mean 7780.29
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.3591, Regression, Linear; Mean Difference (Final Values) = -3782.54, 95% CI 2-sided [-12035.72 to 4470.64], Standard Error of Mean 4073.25

7. Primary Outcome: Change in Inflammatory Biomarker Levels: Interferon-gamma (INF-g)
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on INF-g,, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
pg/mL | -0.03 (2.25) | 0.04 (0.95) | -1.09 (1.09)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.9767, Regression, Linear; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-5.22 to 5.07], Standard Error of Mean 2.54
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.3205, Regression, Linear; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-3.29 to 1.11], Standard Error of Mean 1.09

8. Primary Outcome: Change in Inflammatory Biomarker Levels: Monocyte Chemoattractant Protein-1 (MCP-1)
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on MCP-1, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
pg/mL | -14.66 (15.51) | 0.13 (12.09) | -7.24 (11.47)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.4632, Regression, Linear; Mean Difference (Final Values) = -14.79, 95% CI 2-sided [-55.19 to 25.61], Standard Error of Mean 19.96
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.5316, Regression, Linear; Mean Difference (Final Values) = -7.24, 95% CI 2-sided [-30.47 to 15.99], Standard Error of Mean 11.47

9. Primary Outcome: Change in Inflammatory Biomarker Levels: Tumor Necrosis Factor-alpha (TNF-a)
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on TNF-a, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
pg/mL | -0.22 (0.51) | 0.68 (0.44) | -0.67 (0.34)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.1928, Regression, Linear; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-2.27 to 0.47], Standard Error of Mean 0.68
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.0580, Regression, Linear; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.36 to 0.02], Standard Error of Mean 0.34

10. Primary Outcome: Change in Inflammatory Biomarker Levels: GlycA
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on GlycA, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
umol/L | -0.70 (7.42) | 3.44 (8.76) | -8.35 (8.41)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.7185, Regression, Linear; Mean Difference (Final Values) = -4.14, 95% CI 2-sided [-27.24 to 18.96], Standard Error of Mean 11.41
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.3271, Regression, Linear; Mean Difference (Final Values) = -8.35, 95% CI 2-sided [-25.40 to 8.69], Standard Error of Mean 8.41

11. Primary Outcome: Change in Inflammatory Biomarker Levels: Interleukin (IL)-1b
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on IL-1b, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
pg/mL | 0.07 (0.38) | 0.60 (0.34) | -0.31 (0.11)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.3124, Regression, Linear; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.56 to 0.51], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.0106, Regression, Linear; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.54 to -0.08], Standard Error of Mean 0.11

12. Primary Outcome: Change in Inflammatory Biomarker Levels: IL-2ra
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on IL-2ra, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
ng/mL | -79.07 (28.51) | -8.31 (15.48) | 71.72 (132.87)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0408, Regression, Linear; Mean Difference (Final Values) = -70.76, 95% CI 2-sided [-138.42 to -3.11], Standard Error of Mean 33.42
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.5926, Regression, Linear; Mean Difference (Final Values) = 71.72, 95% CI 2-sided [-197.50 to 340.93], Standard Error of Mean 132.87

13. Primary Outcome: Change in Inflammatory Biomarker Levels: IL-12/23
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on IL-12/23, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
pg/mL | 196.84 (43.59) | 5.35 (4.63) | 171.21 (20.30)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0002, Regression, Linear; Mean Difference (Final Values) = 191.49, 95% CI 2-sided [98.18 to 284.81], Standard Error of Mean 46.10
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p < 0.0001, Regression, Linear; Mean Difference (Final Values) = 171.21, 95% CI 2-sided [130.08 to 212.34], Standard Error of Mean 20.30

14. Primary Outcome: Change in Inflammatory Biomarker Levels: IL-17a
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on IL-17a, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
pg/mL | -1.46 (0.39) | 1.17 (0.94) | -1.15 (0.32)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0110, Regression, Linear; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-4.62 to -0.64], Standard Error of Mean 0.98
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.0008, Regression, Linear; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.79 to -0.51], Standard Error of Mean 0.32

15. Primary Outcome: Change in Inflammatory Biomarker Levels: IL-18
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on IL-18, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
pg/mL | 301.21 (483.77) | 456.52 (487.49) | -407.43 (180.70)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.8227, Regression, Linear; Mean Difference (Final Values) = -155.31, 95% CI 2-sided [-1548.66 to 1238.04], Standard Error of Mean 688.28
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.0302, Regression, Linear; Mean Difference (Final Values) = -407.43, 95% CI 2-sided [-773.57 to -41.29], Standard Error of Mean 180.70

16. Primary Outcome: Change in Inflammatory Biomarker Levels: IL-6
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on IL-6, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
pg/mL | -0.45 (0.22) | 0.02 (0.33) | -0.38 (0.21)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.2333, Regression, Linear; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.25 to 0.32], Standard Error of Mean -0.47
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.0713, Regression, Linear; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.80 to 0.03], Standard Error of Mean 0.21

17. Primary Outcome: Change in Inflammatory Biomarker Levels: IL-8
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on IL-8, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
pg/mL | 2.46 (3.35) | 19.33 (16.02) | -2.23 (1.71)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.2869, Regression, Linear; Mean Difference (Final Values) = -16.87, 95% CI 2-sided [-48.48 to 14.75], Standard Error of Mean 15.62
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.1988, Regression, Linear; Mean Difference (Final Values) = -2.23, 95% CI 2-sided [-5.69 to 1.22], Standard Error of Mean 1.71

18. Primary Outcome: Change in Lipid Biomarker Levels: Triglycerides
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Triglycerides, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
mg/dL | 0.48 (9.42) | -1.58 (8.70) | 10.55 (8.26)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.8744, Regression, Linear; Mean Difference (Final Values) = 2.06, 95% CI 2-sided [-24.09 to 28.20], Standard Error of Mean 12.91
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.2093, Regression, Linear; Mean Difference (Final Values) = 10.55, 95% CI 2-sided [-6.18 to 27.29], Standard Error of Mean 8.26

19. Primary Outcome: Change in Lipid Biomarker Levels: Total Cholesterol
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Total cholesterol, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
mg/dL | 12.57 (5.04) | -6.63 (5.45) | -0.79 (4.14)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0135, Regression, Linear; Mean Difference (Final Values) = 19.20, 95% CI 2-sided [4.21 to 34.20], Standard Error of Mean 7.41
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.8499, Regression, Linear; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-9.19 to 7.61], Standard Error of Mean 4.14

20. Primary Outcome: Change in Lipid Biomarker Levels: High-density Lipoprotein (HDL) Cholesterol
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on HDL cholesterol, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
mg/dL | 2.24 (1.31) | -1.42 (1.46) | 1.92 (1.42)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0693, Regression, Linear; Mean Difference (Final Values) = 3.66, 95% CI 2-sided [-0.30 to 7.62], Standard Error of Mean 1.96
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.1841, Regression, Linear; Mean Difference (Final Values) = 1.92, 95% CI 2-sided [-0.96 to 4.80], Standard Error of Mean 1.42

21. Primary Outcome: Change in Lipid Biomarker Levels: HDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on HDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | -0.02 (0.69) | -1.27 (0.77) | 0.91 (0.72)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.2305, Regression, Linear; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [-0.83 to 3.34], Standard Error of Mean 1.03
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.2189, Regression, Linear; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [-0.53 to 2.37], Standard Error of Mean 0.72

22. Primary Outcome: Change in Lipid Biomarker Levels: HDL Particle Size
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on HDL particle size, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nm
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nm | 0.08 (0.05) | 0.19 (0.10) | 0.17 (0.07)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.3212, Regression, Linear; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.34 to 0.11], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.0137, Regression, Linear; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.04 to 0.31], Standard Error of Mean 0.07

23. Primary Outcome: Change in Lipid Biomarker Levels: Large-HDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Large-HDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | 0.46 (0.38) | 0.33 (0.47) | 0.51 (0.36)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.8383, Regression, Linear; Mean Difference (Net) = 0.12, 95% CI 2-sided [-1.09 to 1.33], Standard Error of Mean 0.60
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.1651, Regression, Logistic; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.22 to 1.24], Standard Error of Mean 0.36

24. Primary Outcome: Change in Lipid Biomarker Levels: Small-HDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Small-HDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | -0.02 (1.15) | -2.52 (1.25) | 0.21 (0.84)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.1502, Regression, Linear; Mean Difference (Final Values) = 2.49, 95% CI 2-sided [-0.94 to 5.93], Standard Error of Mean 1.70
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.8054, Regression, Linear; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-1.49 to 1.91], Standard Error of Mean 0.84

25. Primary Outcome: Change in Lipid Biomarker Levels: Medium-HDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Medium-HDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | -0.56 (1.21) | 0.81 (1.17) | 0.17 (0.97)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.4235, Regression, Linear; Mean Difference (Final Values) = -1.37, 95% CI 2-sided [-4.79 to 2.05], Standard Error of Mean 1.69
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Comparison during RCT period; Test type: Superiority; p = 0.8653, Regression, Linear; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-1.80 to 2.13], Standard Error of Mean 0.97

26. Primary Outcome: Change in Lipid Biomarker Levels: Large Medium-HDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Large medium-HDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | 0.02 (1.26) | 1.14 (1.43) | 0.77 (1.00)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.5580, Regression, Linear; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-4.95 to 2.71], Standard Error of Mean 1.89
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.4454, Regression, Linear; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [-1.25 to 2.80], Standard Error of Mean 1.00

27. Primary Outcome: Change in Lipid Biomarker Levels: Low-density Lipoprotein (LDL) Cholesterol
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on LDL cholesterol, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
mg/dL | 12.52 (4.21) | -8.84 (5.25) | -2.92 (4.07)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0027, Regression, Linear; Mean Difference (Final Values) = 21.37, 95% CI 2-sided [7.86 to 34.87], Standard Error of Mean 6.67
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.4775, Regression, Linear; Mean Difference (Final Values) = -2.92, 95% CI 2-sided [-11.17 to 5.33], Standard Error of Mean 4.07

28. Primary Outcome: Change in Lipid Biomarker Levels: LDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on LDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | 112.67 (46.44) | -118.11 (52.45) | -31.89 (41.71)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0021, Regression, Linear; Mean Difference (Final Values) = 230.77, 95% CI 2-sided [89.47 to 372.08], Standard Error of Mean 69.80
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.4493, Regression, Linear; Mean Difference (Final Values) = -31.89, 95% CI 2-sided [-116.40 to 52.61], Standard Error of Mean 41.71

29. Primary Outcome: Change in Lipid Biomarker Levels: LDL Particle Size
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on LDL particle size, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | 0.20 (0.11) | 0.15 (0.13) | 0.03 (0.11)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.8008, Regression, Linear; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.30 to 0.38], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.8068, Regression, Linear; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.19 to 0.24], Standard Error of Mean 0.11

30. Primary Outcome: Change in Lipid Biomarker Levels: Small-LDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Small-LDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | 24.36 (38.72) | -22.61 (40.61) | 4.68 (33.85)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.4079, Regression, Logistic; Mean Difference (Final Values) = 46.96, 95% CI 2-sided [-66.65 to 160.57], Standard Error of Mean 56.12
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.8907, Regression, Linear; Mean Difference (Final Values) = 4.68, 95% CI 2-sided [-63.91 to 73.28], Standard Error of Mean 33.85

31. Primary Outcome: Change in Lipid Biomarker Levels: Large-LDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Large-LDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | 28.95 (26.87) | 21.95 (41.87) | -24.76 (32.59)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.8866, Regression, Linear; Mean Difference (Final Values) = 7.01, 95% CI 2-sided [-91.80 to 105.81], Standard Error of Mean 48.81
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.4527, Regression, Linear; Mean Difference (Final Values) = -24.74, 95% CI 2-sided [-90.78 to 41.30], Standard Error of Mean 32.59

32. Primary Outcome: Change in Lipid Biomarker Levels: Very Large-LDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Very large-LDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | 93.95 (45.38) | -100.74 (48.29) | -29.16 (38.01)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0056, Regression, Linear; Mean Difference (Final Values) = 194.69, 95% CI 2-sided [60.61 to 328.77], Standard Error of Mean 66.23
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.4478, Regression, Linear; Mean Difference (Final Values) = -29.16, 95% CI 2-sided [-106.17 to 47.85], Standard Error of Mean 38.01

33. Primary Outcome: Change in Lipid Biomarker Levels: Very Low-density Lipoprotein (VLDL) Particle Size
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on VLDL particle size, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | 3.19 (2.19) | 0.04 (1.69) | 1.50 (1.41)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.2704, Regression, Linear; Mean Difference (Final Values) = 3.14, 95% CI 2-sided [-2.55 to 8.83], Standard Error of Mean 2.81
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.2950, Regression, Linear; Mean Difference (Final Values) = 1.50, 95% CI 2-sided [-1.36 to 4.36], Standard Error of Mean 1.41

34. Primary Outcome: Change in Lipid Biomarker Levels: VLDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on VLDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | -9.32 (4.85) | 7.42 (4.34) | -0.11 (3.37)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0149, Regression, Linear; Mean Difference (Final Values) = -16.74, 95% CI 2-sided [-30.03 to -3.45], Standard Error of Mean 6.57
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.9734, Regression, Linear; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-6.93 to 6.71], Standard Error of Mean 3.37

35. Primary Outcome: Change in Lipid Biomarker Levels: VLDL Triglycerides
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on VLDL triglycerides, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
mg/dL | -4.88 (8.85) | 4.33 (7.57) | 11.14 (7.33)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.4384, Regression, Linear; Mean Difference (Net) = -9.21, 95% CI 2-sided [-33.03 to 14.60], Standard Error of Mean 11.76
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.1373, Regression, Linear; Mean Difference (Final Values) = 11.14, 95% CI 2-sided [-3.72 to 25.99], Standard Error of Mean 7.33

36. Primary Outcome: Change in Lipid Biomarker Levels: Small-VLDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Small-VLDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | -5.84 (2.72) | 9.87 (5.27) | -0.50 (2.07)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0097, Regression, Linear; Mean Difference (Final Values) = -15.71, 95% CI 2-sided [-27.39 to -4.03], Standard Error of Mean 5.77
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.8119, Regression, Linear; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-4.69 to 3.70], Standard Error of Mean 2.07

37. Primary Outcome: Change in Lipid Biomarker Levels: Medium-VLDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Medium-VLDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | -3.50 (2.98) | -3.84 (3.50) | -1.86 (2.43)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.9415, Regression, Linear; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-8.91 to 9.59], Standard Error of Mean 4.57
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.4485, Regression, Linear; Mean Difference (Final Values) = -1.86, 95% CI 2-sided [-6.77 to 3.06], Standard Error of Mean 2.43

38. Primary Outcome: Change in Lipid Biomarker Levels: Large Medium-VLDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Large medium-VLDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | -2.89 (3.33) | -2.97 (3.98) | 0.38 (2.59)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.9880, Regression, Linear; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-10.37 to 10.53], Standard Error of Mean 5.16
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.8836, Regression, Linear; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-4.86 to 5.63], Standard Error of Mean 2.59

39. Primary Outcome: Change in Lipid Biomarker Levels: Large-VLDL Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Large-VLDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | 0.29 (0.86) | 0.57 (0.99) | 2.30 (1.08)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.8321, Regression, Linear; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-2.91 to 2.36], Standard Error of Mean 1.30
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.0394, Regression, Linear; Mean Difference (Final Values) = 2.30, 95% CI 2-sided [0.12 to 4.48], Standard Error of Mean 1.08

40. Primary Outcome: Change in Lipid Biomarker Levels: Intermediate-density Lipoprotein (IDL) Particle Number
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on IDL particle number, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
nmol/L | 50.86 (25.89) | -101.79 (36.04) | -2.97 (25.70)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.0012, Regression, Linear; Mean Difference (Final Values) = 152.68, 95% CI 2-sided [64.07 to 241.23], Standard Error of Mean 43.76
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.9085, Regression, Linear; Mean Difference (Final Values) = -2.97, 95% CI 2-sided [-55.04 to 49.09], Standard Error of Mean 25.70

41. Primary Outcome: Change in Lipid Biomarker Levels: Cholesterol Efflux Capacity
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Cholesterol efflux capacity, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
  The ability to promote cholesterol efflux from macrophages is a classic function of HDL that is thought to be an important mechanism by which HDL protects against atherosclerosis. HDL cholesterol efflux capacity assays are performed based on published methods using J774 cells derived from a murine macrophage cell line (Mehta NN Atherosclerosis 2012). Efflux is calculated as a unitless measure by using the following formula: [(µCi of 3H-cholesterol in media containing apoB-depleted subject plasma - µCi of 3H-cholesterol in plasma-free media) / (µCi of 3H-cholesterol in media containing apoB-depleted pooled control plasma-µCi of 3H-cholesterol in pooled control plasma-free media)].
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: unitless (see description)
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
unitless (see description) | 0.09 (0.03) | 0.03 (0.03) | 0.04 (0.03)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.1792, Regression, Linear; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.03 to 0.14], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.2559, Regression, Linear; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.03 to 0.10], Standard Error of Mean 0.03

42. Primary Outcome: Change in Lipid Biomarker Levels: Apolipoprotein-B
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Apolipoprotein-B, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
ug/mL | 0.11 (0.09) | -0.04 (0.09) | 0.10 (0.06)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Test type: Superiority; p = 0.2453, Regression, Linear; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.11 to 0.41], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.1087, Regression, Linear; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.02 to 0.23], Standard Error of Mean 0.06

43. Primary Outcome: Change in Lipid Biomarker Levels: Fetuin-A
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Fetuin-A, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
ug/mL | 10.22 (29.47) | -38.21 (56.05) | -49.56 (27.84)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.4368, Regression, Linear; Mean Difference (Final Values) = 48.43, 95% CI 2-sided [-76.31 to 173.16], Standard Error of Mean 61.62
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.0833, Regression, Linear; Mean Difference (Final Values) = -49.56, 95% CI 2-sided [-105.97 to 6.85], Standard Error of Mean 27.84

44. Primary Outcome: Change in Metabolic Biomarker Levels: Adiponectin
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Adiponectin, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
ug/mL | 0.04 (0.79) | 0.32 (0.77) | 0.38 (0.51)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.8036, Regression, Linear; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-2.52 to 1.97], Standard Error of Mean 1.11
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.4608, Regression, Linear; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.65 to 1.40], Standard Error of Mean 0.51

45. Primary Outcome: Change in Metabolic Biomarker Levels: Leptin
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Leptin, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
pg/mL | 8022.19 (2576.52) | 4701.61 (2184.57) | 6926.25 (2257.84)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.3370, Regression, Linear; Mean Difference (Final Values) = 3320.58, 95% CI 2-sided [-3592.52 to 10233.67], Standard Error of Mean 3414.90
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.0040, Regression, Linear; Mean Difference (Final Values) = 6926.25, 95% CI 2-sided [2351.43 to 11501.07], Standard Error of Mean 2257.84

46. Primary Outcome: Change in Metabolic Biomarker Levels: Insulin
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Insulin, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
pg/mL | 36.19 (116.40) | 105.13 (51.42) | -7.96 (85.98)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.6042, Regression, Linear; Mean Difference (Final Values) = -68.95, 95% CI 2-sided [-335.97 to 198.08], Standard Error of Mean 131.90
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.9267, Regression, Linear; Mean Difference (Final Values) = -7.96, 95% CI 2-sided [-182.18 to 166.26], Standard Error of Mean 85.98

47. Primary Outcome: Change in Metabolic Biomarker Levels: Glucose
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on Glucose, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 22 | 19 | 39
mg/dL | 2.41 (3.34) | -1.79 (4.02) | 3.41 (3.43)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.4226, Regression, Linear; Mean Difference (Final Values) = 4.20, 95% CI 2-sided [-6.28 to 14.68], Standard Error of Mean 5.18
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.3270, Regression, Linear; Mean Difference (Final Values) = 3.41, 95% CI 2-sided [-3.54 to 10.36], Standard Error of Mean 3.43

48. Primary Outcome: Change in Metabolic Biomarker Levels: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on HOMA-IR, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
  HOMA-IR, a method used to quantify insulin resistance and beta-cell function, is expressed using fasting blood glucose and insulin levels. It is calculated using the formula (HOMA-IR = fasting glucose [mg/dl] * fasting insulin [mU/ml]/405).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: unitless (see description)
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 19 | 38
unitless (see description) | 0.07 (1.37) | 0.55 (0.49) | -0.07 (0.89)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period; Test type: Superiority; p = 0.7507, Regression, Linear; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-3.56 to 2.59], Standard Error of Mean 1.52
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Global change from baseline after 52 weeks of active treatment; Test type: Superiority; p = 0.9348, Regression, Linear; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-1.88 to 1.73], Standard Error of Mean 0.89

49. Secondary Outcome: Number of Participants Achieving PASI75 (75% or Greater Reduction in PASI Score)
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on PASI75, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
  Binary measure of change in psoriasis activity; 75% or greater reduction in PASI score compared to baseline.
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Measure: Count of Participants; unit: Participants
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 22 | 19 | 39
Participants | 17 | 2 | 28
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Test type: Superiority; p = 0.0005, Chi-squared; Difference of proportions = 0.67, 95% CI 2-sided [0.45 to 0.89]
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Test type: Other — 95% CI of proportion achieving PASI75 at end of study; Proportion = 0.72, 95% CI 2-sided [0.55 to 0.85]

50. Secondary Outcome: Number of Participants Achieving PASI90 (90% or Greater Reduction in PASI Score)
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on PASI90, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
  Binary measure of change in psoriasis activity; 90% or greater reduction in PASI score compared to baseline.
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Measure: Count of Participants; unit: Participants
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 22 | 19 | 39
Participants | 9 | 0 | 19
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Test type: Superiority; p = 0.0016, Chi-squared; Difference of proportions = 0.41, 95% CI 2-sided [0.20 to 0.62]
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Test type: Other — 95% CI of proportion achieving PASI90 at end of study; Proportion = 0.49, 95% CI 2-sided [0.32 to 0.65]

51. Secondary Outcome: Number of Participants Achieving Physician Global Assessment (PGA) Clear/Almost Clear
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on PGA clear/almost clear, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
  Binary measure of psoriasis disease activity at measurement time points; Physician Global Assessment score <1.5 (clear/almost clear)
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Measure: Count of Participants; unit: Participants
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 22 | 19 | 39
Participants | 14 | 2 | 18
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Comparison during RCT period for binary Physician Global Assessment; Test type: Superiority; p = 0.0005, Chi-squared; Difference of proportions = 0.53, 95% CI 2-sided [0.29 to 0.78]
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Test type: Other — 95% CI of proportion achieving PGA clear/almost clear at end of study; Proportion = 0.46, 95% CI 2-sided [0.30 to 0.63]

52. Secondary Outcome: Change in Patient-Reported Outcomes: MEDFICTS
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on MEDFICTS, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
  MEDFICTS (Meats, Eggs, Dairy, Fried foods, fat In baked goods, Convenience foods, fats added at the Table, and Snacks), a brief dietary assessment instrument, has been provided as part of the National Cholesterol Education Program (NCEP) Adult Treatment Panel (ATP) guidelines as a free tool to use for proper cardiovascular diet assessment. The questionnaire yields a continuous score (ranging from 0 to 216), with a score of <40 indicating adherence to the Therapeutic Lifestyle Changes (TLC) diet (intake of <7% of energy from saturated fat, <30% of energy from total fat, and <200 mg dietary cholesterol/day).
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Measure: Mean (Standard Error); unit: MEDFICTS score
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 22 | 19 | 41
MEDFICTS score | -5.68 (3.97) | -14.00 (4.98) | 8.32 (6.30)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Test type: Superiority; p = 0.1944, Regression, Linear; Mean Difference (Final Values) = 8.32, 95% CI 2-sided [-4.42 to 21.06], Standard Error of Mean 6.30
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Test type: Superiority; p = 0.0011, Regression, Linear; Mean Difference (Final Values) = -12.33, 95% CI 2-sided [-19.40 to -5.25], Standard Error of Mean 3.50

53. Secondary Outcome: Change in Patient-reported Physical Activity Assessments: IPAQ
Description: To assess the effects of ustekinumab, as compared to placebo, at Week 12 (RCT period) in patients with moderate to severe psoriasis on IPAQ, and assess global change at end study (Week 52 for Ustekinumab arm, Week 64 for Placebo arm; active treatment period).
  IPAQ is an instrument designed primarily for population surveillance of physical activity among adults with activity measured in metabolic equivalent (MET)-minutes per week.
Time Frame: Baseline - Week 12; Baseline - End of Study Visit (Week 52 or Week 64)
Measure: Mean (Standard Error); unit: MET-minutes/week
Arm/Group | Ustekinumab (RCT Period) | Placebo (RCT Period) | Total (Active Treatment Period)
Number analyzed (Participants) | 21 | 16 | 37
MET-minutes/week | 73.69 (808.45) | 853.28 (562.37) | -779.59 (1049.99)
Statistical Analysis 1: Comparison: Ustekinumab (RCT Period) vs Placebo (RCT Period); Test type: Superiority; p = 0.4628, Regression, Linear; Mean Difference (Final Values) = -779.59, 95% CI 2-sided [-2911.19 to 1352.01], Standard Error of Mean 1049.99
Statistical Analysis 2: Comparison: Total (Active Treatment Period); Test type: Superiority; p = 0.2209, Regression, Linear; Mean Difference (Final Values) = -910.84, 95% CI 2-sided [-2395.95 to 574.27], Standard Error of Mean 729.96

ADVERSE EVENTS:
Time Frame: 52 weeks for Ustekinumab arm, 64 weeks for Placebo arm.
Description: For each subject, AEs and SAEs occurring after informed consent is obtained should be recorded until the subject has completed his/her participation in the study.
  A serious adverse event must be reported if it occurs during a subject's participation in the Study (whether receiving Study Product or not) and within 12 weeks of receiving the last dose of Study Product in a clinical trial, whichever is longer.
Groups:
- Ustekinumab (Stelara): Ustekinumab (Stelara) subcutaneous injection 45mg (if person's weight is 100kg or less) or 90mg (if person's weight is greater than 100kg) at day 0 and week 4 followed by every 12-week dosing thereafter. From Baseline to Week 52.
- Placebo (RCT Period): Placebo subcutaneous injection will be given according to the same dose and schedule as the active comparator. From Baseline to Week 12 (RCT period only).
- Placebo (Active Treatment Period): Placebo arm after crossing over to receive ustekinumab, following the same dosing schedule of the Ustekinumab arm. From Week 12 to Week 64 (52 weeks of active treatment period).
Arm/Group | Ustekinumab (Stelara) | Placebo (RCT Period) | Placebo (Active Treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 3/19
Other Adverse Events (participants affected / at risk) | 14/22 | 3/21 | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ustekinumab (Stelara) (N=22) | Placebo (RCT Period) (N=21) | Placebo (Active Treatment Period) (N=19)
Endometritis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vasovagal reaction (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ustekinumab (Stelara) (N=22) | Placebo (RCT Period) (N=21) | Placebo (Active Treatment Period) (N=19)
Allergies to foods, food additives, drugs and other chemicals (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Common cold (Infections and infestations) | 6 (6) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pain/Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 11 (11) | 3 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Alkaline Phosphatase Increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anhedonia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Blistering (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Irritant Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dysplastic Nevus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ear And Labyrinth Disorders/Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic Lesion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Latent Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rash/Rash Acneiform/Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (General disorders) | 1 (1) | 0 (0) | 1 (1)
Trichomoniasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Uterine Fibroids Enlarged (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Would Healing Delayed (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT02187172/Prot_SAP_000.pdf